CLINICAL TRIAL: NCT07005349
Title: Rule of THUMB: A Multi-centre Cluster Trial Evaluating the Implementation of a Perioperative Care Complex Intervention to Improve Outcomes From Haemorrhage During and After Caesarean Section in African Hospitals
Brief Title: THUMB: Multi-centre Cluster Trial for Caesarean Section Haemorrhage
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bruce Biccard (Other)
Responsible Party: Sponsor-Investigator, Bruce Biccard, Chief Investigator, University of Cape Town
Organization: University of Cape Town (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: The Rule of THUMB trial
Record Dates: First submitted 2025-04-14; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control phase (No Intervention): Control data will be collected at all hospitals over a two-week period (usual care phase). Patients in the control phase will receive the current standard postoperative care.
- Intervention (Active Comparator): The intervention (a quality improvement programme) will then be implemented by the unit for all patients, aimed at delivering care that is already known to be effective in delivering better patient outcomes.
  Interventions: Other: Quality improvement program

INTERVENTIONS:
Other: Quality improvement program — The intervention comprises two mandatory risk assessments (preoperatively in theatre and postoperatively prior to discharge from the recovery area) which are linked to hospital-specific responses. Assessments for bleeding will occur intraoperatively (through direct vision, haemodynamic changes and/or measurement of blood loss) and postoperatively (with the use of the rapid assessment tool). If bleeding is diagnosed at any point, the THUMB checklist will be used to activate bundled care. On discharge from recovery, high-risk patients will be scheduled to receive a postoperative ward visit within four hours, when a further assessment for bleeding will occur.
  Arms: Intervention

SUMMARY:
The quality improvement project evaluating the delivery of a perioperative care complex intervention to improve haemorrhage-related outcomes in patients undergoing caesarean section. The objectives of the current study will be:

1. To evaluate whether implementation of the 'Rule of THUMB' perioperative complex intervention increases risk assessment, diagnosis and compliance with proven interventions for haemorrhage during and after caesarean section.
2. To understand the influence of contextual and socio-dynamic factors on how the trial results were achieved and how the intervention mechanisms did, or did not, work in practice (the process evaluation). The findings from this study will be used subsequently to modify and improve the quality improvement intervention, so that it can be delivered at scale across Africa and assess its impact on haemorrhage during and after caesarean section in the future.

DETAILED DESCRIPTION:
The study involves a complex intervention to improve maternal outcomes for patients undergoing caesarean section based on early diagnosis of haemorrhage during and after surgery coupled to early treatment through first-responder protocolised treatment using a care bundle of five elements called the rule of THUMB. The intervention is essentially a quality improvement programme aimed at delivering better care, care that is already known to be effective in delivering better patient outcomes. The intervention comprises two mandatory risk assessments (preoperatively in theatre and postoperatively prior to discharge from the recovery area) which are linked to hospital-specific responses. Assessments for bleeding will occur intraoperatively (through direct vision, haemodynamic changes and/or measurement of blood loss) and postoperatively (with the use of the rapid assessment tool). If bleeding is diagnosed at any point, the THUMB checklist will be used to activate bundled care. On discharge from recovery, high-risk patients will be scheduled to receive a postoperative ward visit within four hours, when a further assessment for bleeding will occur. Staff at each hospital will collect data for the two-week usual care (control) phase describing usual perioperative care. This will be followed by a period of co-design and training (2-6 weeks, as required), and then implementation of the intervention phase for a further two weeks at each hospital. The initial intervention will be modified in accordance with data collected during the usual care phase, in conjunction with local stakeholders. Further intervention refinement will occur after each period of data recruitment and analysis. Two intervention cycles will occur. The intervention is essentially a quality improvement programme aimed at delivering better care, care that is already known to be effective in delivering better patient outcomes. The intervention aims to improve compliance with recommended care for prevention and treatment of haemorrhage during and after caesarean section by creating a bundle of care that is delivered simultaneously (not sequentially) by first responders. It includes two mandated risk assessments before and after surgery, and implementation of the THUMB care bundle either in response to bleeding intraoperatively or in recovery or the ward through the rapid assessment tool.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who requires a caesarean section in participating countries with hospitals that routinely perform caesarean section.

Exclusion Criteria:

* Patients who opt out of the trial will be excluded.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 2400 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Patient assessed as high-risk for postpartum haemorrhage | 6 months
  To evaluate the effect of the trial intervention on identification of high-risk patients
Administration of uterotonics intra- or postoperatively | 6 months
  To evaluate the effect of the trial intervention on administration of uterotonics
Administration of tranexamic acid intra- or postoperatively | 6 months
  To evaluate the effect of the trial intervention on administration of tranexamic acid
Uterine massage intra- or postoperatively after delivery of the baby | 6 months
  To evaluate the effect of the trial intervention on uterine massage
A postoperative clinician visit within four hours of discharge to the ward | 6 months
  To evaluate the effect of the trial intervention on clinician ward visit postoperatively

SECONDARY OUTCOMES:
Diagnosis of postpartum haemorrhage | 6 months
  To evaluate the effect of the trial intervention on a diagnosis of postpartum haemorrhage
30 day in-hospital mortality | 6 months
  To evaluate the effect of the trial intervention on 30 day in-hospital mortality
Repeat laparotomy for suspected haemorrhage | 6 months
  To evaluate the effect of the trial intervention on repeat laparotomy for suspected haemorrhage
Duration of hospital stay | 6 months
  To evaluate the effect of the trial intervention on duration of hospital stay
Referral to higher level of care for further management of bleeding/resuscitation | 6 months
  To evaluate the effect of the trial intervention on referral to higher level of care for further management of bleeding/resuscitation

CONTACTS AND LOCATIONS:
Overall Officials: BRUCE BICCARD, PhD, Principal Investigator — University of Cape Town

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with researchers upon request, including, the supporting information selected below.
Supporting Information: Study Protocol, SAP
Time Frame: Following publication of the results, IPD will be made available upon request.
Access Criteria: Any researchers, and clinicians or healthcare workers continuing care of the participants after the study, as well as the participants themselves.

REFERENCES:
- [Result] Sobhy S, Arroyo-Manzano D, Murugesu N, Karthikeyan G, Kumar V, Kaur I, Fernandez E, Gundabattula SR, Betran AP, Khan K, Zamora J, Thangaratinam S. Maternal and perinatal mortality and complications associated with caesarean section in low-income and middle-income countries: a systematic review and meta-analysis. Lancet. 2019 May 11;393(10184):1973-1982. doi: 10.1016/S0140-6736(18)32386-9. Epub 2019 Mar 28. PMID 30929893
- [Result] Bishop D, Dyer RA, Maswime S, Rodseth RN, van Dyk D, Kluyts HL, Tumukunde JT, Madzimbamuto FD, Elkhogia AM, Ndonga AKN, Ngumi ZWW, Omigbodun AO, Amanor-Boadu SD, Zoumenou E, Basenero A, Munlemvo DM, Youssouf C, Ndayisaba G, Antwi-Kusi A, Gobin V, Forget P, Mbwele B, Ndasi H, Rakotoarison SR, Samateh AL, Mehyaoui R, Patel-Mujajati U, Sani CM, Esterhuizen TM, Madiba TE, Pearse RM, Biccard BM; ASOS investigators. Maternal and neonatal outcomes after caesarean delivery in the African Surgical Outcomes Study: a 7-day prospective observational cohort study. Lancet Glob Health. 2019 Apr;7(4):e513-e522. doi: 10.1016/S2214-109X(19)30036-1. PMID 30879511
- [Result] Sheldon WR, Blum J, Vogel JP, Souza JP, Gulmezoglu AM, Winikoff B; WHO Multicountry Survey on Maternal and Newborn Health Research Network. Postpartum haemorrhage management, risks, and maternal outcomes: findings from the World Health Organization Multicountry Survey on Maternal and Newborn Health. BJOG. 2014 Mar;121(Suppl 1):5-13. doi: 10.1111/1471-0528.12636. PMID 24641530
- [Result] Gallos I, Devall A, Martin J, Middleton L, Beeson L, Galadanci H, Alwy Al-Beity F, Qureshi Z, Hofmeyr GJ, Moran N, Fawcus S, Sheikh L, Gwako G, Osoti A, Aswat A, Mammoliti KM, Sindhu KN, Podesek M, Horne I, Timms R, Yunas I, Okore J, Singata-Madliki M, Arends E, Wakili AA, Mwampashi A, Nausheen S, Muhammad S, Latthe P, Evans C, Akter S, Forbes G, Lissauer D, Meher S, Weeks A, Shennan A, Ammerdorffer A, Williams E, Roberts T, Widmer M, Oladapo OT, Lorencatto F, Bohren MA, Miller S, Althabe F, Gulmezoglu M, Smith JM, Hemming K, Coomarasamy A. Randomized Trial of Early Detection and Treatment of Postpartum Hemorrhage. N Engl J Med. 2023 Jul 6;389(1):11-21. doi: 10.1056/NEJMoa2303966. Epub 2023 May 9. PMID 37158447
- [Result] APORG Caesarean Delivery Haemorrhage Group. Identifying interventions to reduce peripartum haemorrhage associated with caesarean delivery in Africa: A Delphi consensus study. PLOS Glob Public Health. 2022 Aug 31;2(8):e0000455. doi: 10.1371/journal.pgph.0000455. eCollection 2022. PMID 36962699
- [Result] Althabe F, Therrien MNS, Pingray V, Hermida J, Gulmezoglu AM, Armbruster D, Singh N, Guha M, Garg LF, Souza JP, Smith JM, Winikoff B, Thapa K, Hebert E, Liljestrand J, Downe S, Garcia Elorrio E, Arulkumaran S, Byaruhanga EK, Lissauer DM, Oguttu M, Dumont A, Escobar MF, Fuchtner C, Lumbiganon P, Burke TF, Miller S. Postpartum hemorrhage care bundles to improve adherence to guidelines: A WHO technical consultation. Int J Gynaecol Obstet. 2020 Mar;148(3):290-299. doi: 10.1002/ijgo.13028. Epub 2019 Dec 23. PMID 31709527
- [Result] Seim AR, Alassoum Z, Souley I, Bronzan R, Mounkaila A, Ahmed LA. The effects of a peripartum strategy to prevent and treat primary postpartum haemorrhage at health facilities in Niger: a longitudinal, 72-month study. Lancet Glob Health. 2023 Feb;11(2):e287-e295. doi: 10.1016/S2214-109X(22)00518-6. PMID 36669809
- [Result] Main EK, Goffman D, Scavone BM, Low LK, Bingham D, Fontaine PL, Gorlin JB, Lagrew DC, Levy BS. National Partnership for Maternal Safety: consensus bundle on obstetric hemorrhage. Anesth Analg. 2015 Jul;121(1):142-148. doi: 10.1097/AOG.0000000000000869. PMID 26091046

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-18): https://cdn.clinicaltrials.gov/large-docs/49/NCT07005349/Prot_SAP_000.pdf